CLINICAL TRIAL: NCT06747637
Title: Demonstrating the Efficacy of "Unidos en el Cuidado" (United in Caring): A Spanish-Language Program for Latino Caregivers of Persons Living With Dementia
Brief Title: Demonstrating the Efficacy of a Spanish-Language Program for Latino Dementia Caregivers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: California Department of Public Health (Other)
Responsible Party: Principal Investigator, Maria P. Aranda, Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AWD-00008709
Record Dates: First submitted 2024-12-11; First posted 2024-12-24 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Caregiver Burden of People With Dementia
Keywords: wait list control interventional study

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Treatment Group Receives the Classes Soon after Randomization (Experimental): The Spanish-language caregiver classes are called Unidos en el Cuidado and are taught online by Alzheimer's Los Angeles. Sessions are provided at no cost and held weekly for about 2 hours.
  Interventions: Other: Skill-building classes
- Group B: Wait List Control Group Receives the Classes after a Waiting Period (Active Comparator): This wait list control group receives the same classes but after a 3-4 week waiting period.
  Interventions: Other: Wait list control group

INTERVENTIONS:
Other: Skill-building classes — Unidos en el Cuidado is a manualized, multi-family group intervention provided at no cost vis-à-vis videoconferencing or on-site by trained facilitators Sessions are held weekly for 1.5 hours. Class components include caregiver role identity; skills-building; knowledge attainment; attitudinal changes; resource-sharing; practice/role-plays; homework; videos, handouts. Classes will be provided online with some classes offered in the community, if available
  Arms: Group A: Treatment Group Receives the Classes Soon after Randomization
Other: Wait list control group — The intervention is the same; the wait period is longer to receive the intervention described in Group A.
  Arms: Group B: Wait List Control Group Receives the Classes after a Waiting Period

SUMMARY:
The investigators will test the efficacy of Unidos en el Cuidado® (United in Caring, herein Unidos), a 3-session, culturally-adapted, group psychoeducational and skill-building intervention for 226 Spanish-speaking family caregivers in California.

DETAILED DESCRIPTION:
The investigators will test the efficacy of Unidos en el Cuidado® (United in Caring, herein Unidos), a 3-session, culturally-adapted, group psychoeducational and skill-building intervention for 226 Spanish-speaking family caregivers in California.

Based on a wait list trial design, and 4 observation points (baseline, post-intervention, 3-month and 6-month follow-ups), the investigators propose to demonstrate the efficacy of this new intervention (Aim 1), and evaluate for potential moderating conditions across subgroups (Aim 2; age, gender, educational level, etc.). Based on this quantitative component, the investigators will answer the following two aims:

Aim #1. (Efficacy) Compared to a waitlist control group, is Unidos efficacious with regards to primary outcomes-PHQ-9 depression symptoms, RMBPC reactivity to memory and behavior problems, anxiety symptoms, and secondary outcomes-caregiver mastery, competence, and meaning over time?

Aim #2: (Moderators). Do moderating conditions exist such that the intervention is more or less efficacious for subgroups based on age, gender, PLWD functioning?

Qualitative component: After class completion, the investigators will draw from 40-50 focus group participants to elucidate the satisfaction and acceptability of the program. Both Unidos and wait list control participants will be randomly selected for focus group interviews which will be guided by open-ended inquiries around the nuanced, in-depth perspectives of program participation, acceptability, and recommendations (Aim 3).

Aim #3: (Experience/Satisfaction). Will qualitative reports from focus groups signal satisfaction, nuanced differences with respect to the nature, structure, cultural/ language considerations of Unidos, and recommendations?

Based on the scientific team and community partner's established expertise in dementia care, caregiving services, and underrepresented groups, the project is well positioned to address the linguistic and cultural preferences and needs of diverse Californians and the providers that serve them.

ELIGIBILITY:
Inclusion Criteria:

* identifies with being Hispanic or Latino descent
* speaks and reads Spanish
* dementia family caregivers living (or recently lived) in California or whose care recipient lives (or recently lived) in California
* who identify as women, men, or non-binary,
* age 18 years or older

Exclusion Criteria:

* Severe sensory or physical conditions that interfere with ongoing participation.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2025-06-04 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Depressive symptoms | baseline; post-intervention (within 1 week of completing intervention); 3-months; 6-months from baseline
  Patient Health Questionnaire 9 item standardized scale: min. to max values=0 to 27; higher values indicate worse outcomes
Presence and reaction to memory and behavior problems shown by person with dementia | baseline; post-intervention (within 1 week of completing intervention); 3-months; 6-months from baseline
  Revised Memory and Behavior Problems Checklist standardized scale:
  1. Symptom presence (yes/no); min. to max values=0 to 24; higher values indicate worse outcomes
  2. Symptom reaction: Include only items with frequency scores of 1 to 4 in the reaction scoring. Compute the mean reaction score by summing reaction scores of these items and then dividing by the number of items included in the sum. the range for each subscale is 0 to 4. Higher values indicate worse outcomes
Anxiety symptoms | baseline; post-intervention (within 1 week of completing intervention); 3-months; 6-months from baseline
  Generalized Anxiety Disorder 7 item standardized scale: min. to max values=0 to 24; higher values indicate worse outcomes

SECONDARY OUTCOMES:
Caregiver Mastery | baseline; post-intervention (within 1 week of completing intervention); 3-months; 6-months from baseline
  Caregiver Mastery standardized scale: min. to max values=0 to 12; higher values indicate better outcomes
Caregiver Competence | baseline; post-intervention (within 1 week of completing intervention); 3-months; 6-months from baseline
  Caregiver Competence standardized scale: min. to max values=0 to 12; higher values indicate better outcomes
Caregiver Meaning | baseline; post-intervention (within 1 week of completing intervention); 3-months; 6-months from baseline
  Caregiver Meaning standardized scale: min. to max values=0 to 24; higher values indicate better outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Maria P Aranda, PhD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Griffiths PC, Kovaleva M, Higgins M, Langston AH, Hepburn K. Tele-Savvy: An Online Program for Dementia Caregivers. Am J Alzheimers Dis Other Demen. 2018 Aug;33(5):269-276. doi: 10.1177/1533317518755331. Epub 2018 Mar 16. PMID 29544342